CLINICAL TRIAL: NCT05203718
Title: A Mixed Methods, Single-group, Single-center Feasibility Study of a Food Response Training to Reduce Unhealthy Dietary Intake and Promote Weight Loss in Racially and Ethnically Diverse Patients With Obesity
Brief Title: The Retrain Your Brain for Healthy Eating Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-00889
Record Dates: First submitted 2022-01-20; First posted 2022-01-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Food Response Training (FRT)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with Obesity (Experimental): NYU Langone Health patients ≥18 to 80 years of age with a BMI ≥30.0 kg/m2
  Interventions: Behavioral: Food Response Training (FRT)

INTERVENTIONS:
Behavioral: Food Response Training (FRT) — All patients will complete the 12-week FRT intervention consisting of one in-person session (during the baseline visit) and three weekly sessions at home, one delivered via video conference (WebEx) and two self-guided. Food Response Training (FRT) is a computer-based attention bias modification intervention. The intervention will be delivered on a computer or smart device (e.g. iPhone). Patients will use the FoodTrainer application available for Android and iPhone (https://www.exeter.ac.uk/foodt/about/).

SUMMARY:
The aim of this mixed methods, single-group, single-center study will be to examine the feasibility of a food response training (FRT). This study will be conducted in patients with obesity recruited from NYU Langone Health. Measurements will occur at screening, baseline, and 3 months, for a subgroup of participants for we will collect saliva samples for genetic analysis at baseline assessment (ancillary study).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to 80 years of age
2. BMI ≥30.0 kg/m2
3. access to a computer or an iPhone/iPad or be willing to use a study loaner smart phone

Exclusion Criteria:

1. pregnant or breastfeeding or plan to become pregnant in the next 6 months, or who become pregnant during the study
2. taking any medication that may impact dietary intake and weight:

   a. Immunosuppressants, steroids, medications for weight loss or to manage blood sugars or a psychiatric condition other than anxiety/depression
3. enrolled in another intervention that could influence dietary intake
4. have had bariatric surgery within the past 2 years
5. unwilling to delay bariatric surgery for the next 6 months
6. who have gained or loss more than 5.5 kg in the previous 3 months
7. unable to participate meaningfully in an intervention that involves using software available in English. The reason for this is that the food training apps have not been designed or validated in audio form or in other languages. (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia)
8. institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have limited control over diet), unwilling or inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Rate of Intervention Uptake | Baseline (Day 0)
  This will be reported as the number of participants who are enrolled and assessed for eligibility.
Rate of Intervention Retention | Week 12
  This will be reported as the number of 12-week survey completers / total enrolled participants.
Health Eating Index (HEI-2015) Score | Week 12
  HEI-2015 is a measure of diet quality used to assess how well a set of foods aligns with key recommendations of the Dietary Guidelines for Americans. The total HEI-2015 score for Americans is 59 out of 100; the higher the score, the more the foods align with key recommendations.

SECONDARY OUTCOMES:
Change in Weight (kg) | Baseline, Week 12
Change in Blood Pressure (BP) | Baseline, Week 12
Change in Waist Circumference (cm) | Baseline, Week 12
Change in Hip Circumference (cm) | Baseline, Week 12
Change in Neck Circumference (cm) | Baseline, Week 12
Change in Food Cravings Questionnaire - Trait (FCQ-T) Score | Baseline, Week 12
  FCQ-T measures the frequency and intensity of food craving experiences in general. The questionnaire has 39 items and response categories range from 1 = never to 6 = always. There are no inverted items. Responses to all items are summed up for a total score. Thus, higher scores represent more frequent and intense food cravings.
Change in Yale Food Addiction Scale (YFAS) | Baseline, Week 12
  YFAS is a measure to identify those who are most likely to be exhibiting markers of substance dependence with the consumption of high fat/high sugar foods. The 25 questions are scored with defined cut-offs (0 = question not significantly met, 1 = question criteria met). After computing cut-offs, the questions under each substance dependence criterion are summed. If the score for the criterion is >/= 1, then the criterion has been met and is scored as 1. If the score = 0, then the criteria has not been met. To score the continuous version of the scale, which resembles a symptom count without diagnosis, all of the scores for each criterion are added up. The total score range is 0-7 (0 symptoms to 7 symptoms). The higher the score, the greater the number of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Jay, MD, MS, Principal Investigator — NYU Langone Health; Sandra Wittleder, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Clinical & Translational Science Institute Clinical Research Center (CTSI CRC), New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Sandra.wittleder@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.